CLINICAL TRIAL: NCT03334604
Title: The Effect of a Multispecies Probiotic on Reducing the Incidence of Antibiotic-associated Diarrhoea in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Winclove Probiotics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAD2017
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-01

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: antibiotic-associated diarrhea; probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multispecies probiotic group (Experimental): 175 participants.
  Interventions: Dietary Supplement: Multispecies probiotic
- Control group (Placebo Comparator): 175 participants.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multispecies probiotic — Multispecies probiotic consisting of Bifidobacterium bifidum W23, Bifidobacterium lactis W51, Lactobacillus acidophilus W37, Lactobacillus acidophilus W55, Lactobacillus paracasei W20, Lactobacillus plantarum W62, Lactobacillus rhamnosus W71 and Lactobacillus salivarius W24 at a dose of 5x10^9 Colony Forming Units (CFU), twice daily, orally.
  Arms: Multispecies probiotic group
Other: Placebo — Placebo identical in taste, smell and color to the multispecies probiotic.
  Arms: Control group

SUMMARY:
In this trial, the investigators aim to assess the effectiveness of a multispecies probiotic consisting of 2 strains of Bifidobacterium (B. bifidum W23, B. lactis W51) and 6 strains of Lactobacillus (L. acidophilus W37, L. acidophilus W55, L. paracasei W20, L. plantarum W62, L. rhamnosus W71, and L. salivarius W24) in reducing the risk of antibiotic-associated diarrhoea in a group of children undergoing antibiotic therapy for common infections.

DETAILED DESCRIPTION:
Certain individual probiotic strains have been proven to be effective in reducing the risk of antibiotic-associated diarrhoea (AAD). However, the effects of using multispecies probiotics remain unclear. The investigators aim to assess the effectiveness of a specific multispecies probiotic preparation (Ecologic AAD Kids) in reducing the incidence of AAD in children.

In this trial, a total of 350 children aged 3 months to 18 years, undergoing antibiotic treatment, will be randomly allocated to receive either a multispecies probiotic consisting of 2 strains of Bifidobacterium (B. bifidum W23, B. lactis W51) and 6 strains of Lactobacillus (L. acidophilus W37, L. acidophilus W55, L. paracasei W20, L. plantarum W62, L. rhamnosus W71, and L. salivarius W24) at a total dose of 10^10 colony-forming units daily, or a placebo, from the first day of antibiotic treatment until 7 days after antibiotic cessation. The primary outcome measure will be the incidence of AAD, defined as ≥3 loose or watery stools (a score of A on the Amsterdam Infant Stool Scale for children younger than 1 year and a score of 5-7 on the Bristol Stool Form scale for children older than 1 year) in 24 hours, caused either by Clostridium difficile or of otherwise unexplained aetiology (after testing for common diarrhoeal pathogens), occurring during and/or up to 7 days after the end of the antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* children receiving oral or intravenous antibiotics for common infections, willing and able to start the probiotic intervention within 24 hours after the start of antibiotic intake, receiving broad-spectrum antibiotics (broad-spectrum penicillins, cephalosporins, fluoroquinolones, clindamycin).

Exclusion Criteria:

* prior use of antibiotics within the previous 4 weeks, presence of a severe or generalised infection, history of severe chronic disease (e.g., cancer, inflammatory bowel disease, tuberculosis), critical/life-threatening illness, immunodeficiency, history of pre-existing diarrhoea within the previous 4 weeks, exclusive breastfeeding, allergy or hypersensitivity to any component of the study product, tube-feeding, use of proton-pump inhibitors, laxatives or anti-diarrhoeal drugs, as well as use of a probiotic product containing L rhamnosus GG or S boulardii 14 days before and during the study.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Incidence of antibiotic-associated diarrhea | Up to 7th day after antibiotic cessation.
  Antibiotic-associated diarrhea will be defined as 3 or more loose or watery stools (a score of A on the Amsterdam Infant Stool Scale or 5-7 on the Bristol Stool Form scale) per day in a 24-hour period, caused by C. difficile infection or of otherwise unexplained aetiology after testing for common diarrhoeal pathogens (rotavirus, adenovirus, norovirus, Campylobacter spp., Salmonella spp., Shigella spp., and Yersinia spp.), occurring during the intervention period.

SECONDARY OUTCOMES:
Incidence of antibiotic-associated diarrhea - alternative definition 1 | Up to 7th day after antibiotic cessation.
  ≥3 loose or watery stools per day for a minimum of a 48-hour period caused by C. difficile infection or of otherwise unexplained aetiology.
Incidence of antibiotic-associated diarrhea - alternative definition 2 | Up to 7th day after antibiotic cessation.
  ≥2 loose or watery stools per day for a minimum of a 24-hour period caused by C. difficile infection or of otherwise unexplained aetiology.
Incidence of diarrhea | Up to 7th day after antibiotic cessation.
  ≥3 loose or watery stools per day for a minimum of 24 hours regardless of its aetiology.
Clostridium difficile-associated diarrhea | Up to 7th day after antibiotic cessation.
  ≥3 loose or watery stools per day for a minimum of 24 hours caused by C. difficile confirmed by the presence of toxin-producing C. difficile in stools.
Duration of diarrhea | Up to 7th day after antibiotic cessation.
  Defined as the time until the normalisation of stool consistency according to the Bristol Stoo Form (BSF) or Amsterdam Infant Stool Scale (AISS) - on BSF numbers 1, 2, 3 and 4; on AISS scale, letters B or C, and the presence of normal stools for 48 h.
Discontinuation of the antibiotic treatment due to severity of diarrhoea | Up to 7th day after antibiotic cessation.
Hospitalisation caused by diarrhoea | Up to 7th day after antibiotic cessation.
Need for intravenous rehydration | Up to 7th day after antibiotic cessation.
Adverse events | Up to 7th day after antibiotic cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Łukasik, MD, Principal Investigator — Department of Paediatrics, The Medical University of Warsaw, Poland
Locations (6):
- Netherlands (4):
  - OLVG location West, Amsterdam
  - Amsterdam UMC, location VUmc, Amsterdam
  - OLVG location East, Amsterdam
  - Amsterdam UMC, location AMC, Amsterdam
- Poland (2):
  - Department of Paediatrics, St. Hedwig of Silesia Hospital, Trzebnica, Silesian Voivodeship
  - Department of Paediatrics, The Medical University of Warsaw, Poland, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
The data collected in the course of this study are available from the Principal Investigator upon reasonable request.

REFERENCES:
- [Derived] Dierikx TH, Malinowska AM, Lukasik J, Besseling-van der Vaart I, Belzer C, Szajewska H, de Meij TGJ; Multispecies Probiotic in AAD Study Group. Probiotics and Antibiotic-Induced Microbial Aberrations in Children: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2418129. doi: 10.1001/jamanetworkopen.2024.18129. PMID 38967929
- [Derived] Lukasik J, Dierikx T, Besseling-van der Vaart I, de Meij T, Szajewska H; Multispecies Probiotic in AAD Study Group. Multispecies Probiotic for the Prevention of Antibiotic-Associated Diarrhea in Children: A Randomized Clinical Trial. JAMA Pediatr. 2022 Sep 1;176(9):860-866. doi: 10.1001/jamapediatrics.2022.1973. PMID 35727573
- [Derived] Lukasik J, Szajewska H. Effect of a multispecies probiotic on reducing the incidence of antibiotic-associated diarrhoea in children: a protocol for a randomised controlled trial. BMJ Open. 2018 Jun 4;8(5):e021214. doi: 10.1136/bmjopen-2017-021214. PMID 29866789